CLINICAL TRIAL: NCT02218684
Title: Tolerability and Pharmacokinetics of 80 mg Telmisartan in Combination With 2, 4, or 6 mg Lacidipine. An Open, Single Rising Dose Group Comparison Trial - Placebo Randomised Double Blind in Each Dose Group - in Male Healthy Subjects
Brief Title: Tolerability and Pharmacokinetics of Telmisartan in Combination With Lacidipine in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1173.1
Record Dates: First submitted 2014-08-15; First posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan; lacidipine

ARMS (4):
- Telmisartan + Lacidipine - low dose (Experimental)
  Interventions: Drug: Telmisartan; Drug: Lacidipine
- Telmisartan + Lacidipine - medium dose (Experimental)
  Interventions: Drug: Telmisartan; Drug: Lacidipine
- Telmisartan + Lacidipine - high dose (Experimental)
  Interventions: Drug: Telmisartan; Drug: Lacidipine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan
  Arms: Telmisartan + Lacidipine - high dose; Telmisartan + Lacidipine - low dose; Telmisartan + Lacidipine - medium dose
Drug: Lacidipine
  Arms: Telmisartan + Lacidipine - high dose; Telmisartan + Lacidipine - low dose; Telmisartan + Lacidipine - medium dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The trial objectives were to investigate the tolerability and pharmacokinetics of 80 mg telmisartan and 2, 4 or 6 mg lacidipine administered concurrently.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male caucasian subjects as determined by results of screening
* Written informed consent in accordance with Good Clinical Practice and local legislation given
* Age >= 18 and <= 50 years
* Broca >= -20% and <= + 20%

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and Electrocardiogram (ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurologic disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (<= 1 month prior to administration or during the trial)
* Use of any drugs which might influence the results of the trial (<= 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (<= 2 months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 60g/day)
* Drug abuse
* Blood donation > 100 ml (<= 4 weeks prior to administration or during the trial)
* Excessive physical activities (<= 10 days prior to administration or during the trial)
* Any laboratory value outside the reference range of clinical relevance

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 1998-09; Primary Completion 1998-11 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum measured concentration of the analyte in plasma) | up to 72 hours after drug administration
Number of subjects with adverse events | up to 72 hours after drug administration

SECONDARY OUTCOMES:
AUC (Area under the concentration-time curve of the analyte in plasma) | up to 72 hours after drug administration
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 72 hours after drug administration
CL/F (Apparent clearance of the analyte in plasma following extravascular administration) | up to 72 hours after drug administration
Vz/F (Apparent volume of distribution of the analyte during the terminal phase) | up to 72 hours after drug administration
MRT (Mean residence time of the analyte in the body) | up to 72 hours after drug administration
t½ (Terminal half-life of the analyte in plasma) | up to 72 hours after drug administration
Number of subjects with abnormal changes in laboratory parameters | up to 72 hours after drug administration
Number of subjects with clinically significant changes in vital signs | up to 72 hours after drug administration